CLINICAL TRIAL: NCT06956521
Title: Intra-Arterial Magnesium Therapy After Mechanical Thrombectomy in Acute Ischemic Stroke
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Omar Tanweer, Director of Cerebrovascular and Endovascular Neurosurgery, Baylor College of Medicine
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: H-50731
Record Dates: First submitted 2024-12-02; First posted 2025-05-04 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Acute Ischemic Stroke
Keywords: stroke; magnesium sulfate; neuroprotection
MeSH Terms: conditions — Ischemic Stroke; Stroke | interventions — Magnesium Sulfate

STUDY DESIGN:
Intervention Model Description: This trial will follow a dose escalation paradigm such that patients are sequentially enrolled into 4 groups. The first patients enrolled will be in the first group that receives the lowest dose. If the IA magnesium dose is safe in this group, the next patients will be enrolled in the 2nd group that receives a higher dose, this continuing until the final group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- 0.25g Magnesium Sulfate (Experimental): 0.25g of magnesium sulfate (MgSO4) will be diluted in 0.9% sodium chloride for intra-arterial (IA) administration via the guide catheter already in place in the intracranial internal carotid artery (ICA) on the affected side for MT. The infusion will be administered over 1-2 minutes.
  Interventions: Drug: Magnesium sulfate
- 0.5g Magnesium Sulfate (Experimental): 0.5g of magnesium sulfate (MgSO4) will be diluted in 0.9% sodium chloride for intra-arterial (IA) administration via the guide catheter already in place in the intracranial ICA on the affected side for MT. The infusion will be administered over 1-2 minutes.
  Interventions: Drug: Magnesium sulfate
- 1.0g Magnesium Sulfate (Experimental): 1.0g of magnesium sulfate (MgSO4) will be diluted in 0.9% sodium chloride for intra-arterial (IA) administration via the guide catheter already in place in the intracranial ICA on the affected side for MT. The infusion will be administered over 1-2 minutes.
  Interventions: Drug: Magnesium sulfate
- 1.5g Magnesium Sulfate (Experimental): 1.5g of magnesium sulfate (MgSO4) will be diluted in 0.9% sodium chloride for intra-arterial (IA) administration via the guide catheter already in place in the intracranial ICA on the affected side for MT. The infusion will be administered over 1-2 minutes.
  Interventions: Drug: Magnesium sulfate

INTERVENTIONS:
Drug: Magnesium sulfate — Following MT and IA injection of MgSO4, patients will also receive a continuous infusion of 16g MgSO4 diluted in 240 ml of 0.9% normal saline, infusing at a rate of 10 ml per hour for 24 hours.
  Other Names: MA 135 magnesium sulfate heptahydrate

SUMMARY:
The goal of this Phase I unblinded, dose-escalation trial is to evaluate the safety and tolerability of intra-arterial magnesium sulfate injection after mechanical thrombectomy in patients experiencing acute ischemic stroke. This trial is one of the first trials to look at IA administration of magnesium sulfate into at risk brain tissue in a selective and localized fashion.

DETAILED DESCRIPTION:
Patients meeting inclusion and exclusion criteria will undergo a baseline neurologic assessment and will be enrolled following informed consent. The patient will then be taken to the Interventional Radiology suite where the patient will undergo MT as per the standard of care. Participation in this study will never delay the timely provision of urgent MT to patients.

Additionally, as part of the study procedure, the patient will be assigned to Treatment Group 1,2, 3 or 4 based on the consecutive sampling scheme. The first 6 patients enrolled will be in group 1 and receive the lowest dose of MgSO4 as described below. If the analysis of this group deems this dosage to be safe, the following patients will be enrolled into group 2. The same scheme will be followed until all 4 groups are enrolled.

Patients in all groups will receive IA MgSO4 as follows (investigational):

Patients in each group will receive the specified dose of MgSO4 (listed below) diluted in 0.9% sodium chloride. The infusion of IA MgSO4 will be administered over 1-2 minutes.

Dose Escalation Schedule Group 1 0.25g IA MgSO4 Group 2 0.5g IA MgSO4 Group 3 1g IA MgSO4 Group 4 1.5g IA MgSO4

Given the minimal safety data on IA MgSO4, this dosage regimen was derived from previous IV MgSO4 studies and a singular IA MgSO4 study in a separate population to cautiously investigate the safety and tolerability for IA MgSO4.

Following MT and IA infusion, patients will receive a continuous infusion of IV MgSO4 for 24 hours. The maintenance infusion will contain 16g of MgSO4 diluted in 240 ml of 0.9% normal saline, infused at a rate of 10 ml per hour for 24 hours. Patients will follow the standard of care monitoring for post-MT patients with the addition of monitoring for magnesium toxicity.

All pre and post imaging is standard of care for this procedure, including follow up MRI (or CT if MRI contraindicated).

Following discharge from the hospital, all patients enrolled in the study protocol will be followed up in the clinic at 3 months to evaluate the patient's functional clinical outcome. If for any reason, the patient cannot come back for a follow-up visit, the PI/Co-PI's will contact the patient via phone/email to gather the required data. A minimum of mRS and NIHSS should be gathered for follow-up data.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with acute cerebral ischemia due to ICA or MCA occlusion
2. Major neurologic deficits: 6≤NIHSS≤20,
3. Premorbid mRS 0 or 1, or 2
4. Patient's clinical attending physician plans MT procedure as part of routine clinical care,
5. undergo MT with a TICI 2a or better recanalization,
6. Signed informed consent.

Exclusion Criteria:

1. Positive pregnancy test;
2. those undergoing MT with a TICI <2a revascularization;
3. tandem occlusion of the cervical common or internal carotid artery; and
4. subjects on therapeutic anticoagulation, as it is a relative contraindication to MT, and could be a confounding variable predisposing to intracranial hemorrhage including coagulation disorders, systematic hemorrhagic tendency, thrombocytopenia <80000/mm3;
5. Second or third-degree heart block without a pacemaker in place,
6. Technical inability to navigate micro-catheter to target clot,
7. Patient already enrolled in another experimental treatment trial. Exclusion criteria 1-3 are all contraindications to magnesium therapy,
8. mRS>2 caused by a history of prior stroke,
9. Severe hepatic dysfunction, severe renal dysfunction (<30 mL/min), increase in ALT or AST (more than 2 times of upper limit of normal value), increase in serum creatinine (more than 1.5 times of upper limit of normal value) or requiring dialysis;
10. Unsuitable for this clinical study assessed by researcher. Subjects will not be excluded if they received IV t-PA as standard of care.
11. patient is on neuromuscular blocking agents including depolarizing (succinylcholine) and nondepolarizing subtypes (rocuronium, vecuronium, etc);
12. patient is taking any form of CNS depressant including barbiturates, narcotics, outside the setting of anesthesia or ICU sedation
13. patients taking digoxin or other cardiac glycoside

Ages: 21 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Systemic MgSO4 Concentration | 6 hours post-MT, 24 hours post-MT
Proportion of severe adverse events | 48 hours post-MT
  severe adverse events including femoral artery dissection, local thrombosis, pseudoaneurysm, arteriovenous fistula, neurotoxicity and loss of reflexes due to magnesium, cardiovascular toxicity (arrythmias, severe bradycardia), respiratory depression

SECONDARY OUTCOMES:
Proportion of patients with Modified Rankin Scale (mRS) 0 to 2 | 90 days post-MT
  mRS is a measure of global disability. Total Scale range is 0-6, with lower values indicating better outcomes. mRS </= 2 is considered functional independence based on modified Rankin score.
Modified Rankin Scales (mRS) | 90 days post-MT
  mRS is a measure of global disability. Total Scale range is 0-6, with lower values indicating better outcomes.
  0. No symptoms at all
  1. No significant disability despite symptoms; able to carry out all usual duties and activities
  2. Slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance
  3. Moderate disability; requiring some help, but able to walk without assistance
  4. Moderately severe disability; unable to walk without assistance and unable to attend to own bodily needs without assistance
  5. Severe disability; bedridden, incontinent and requiring constant nursing care and attention
  6. Dead
Decrease in National Institutes of Health Stroke Scale (NIHSS) | 48 hours post-MT
  NIHSS is a measure of neurologic deficit. Total Score range 0-42, with higher scores indicating greater severity. The 11 domains assessed are:
  1a-c Level of consciousness 2. Best Gaze 3. Visual 4. Facial Palsy 5a. Motor left arm 5b. Motor right arm 6a. Motor left leg 6b. Motor right leg 7. Limb Ataxia 8. Sensory 9. Best Language 10. Dysarthria 11. Extinction and Inattention
Proportion of symptomatic intracranial hemorrhage (sICH) | 48 hours post-MT
  sICH defined as 4 or more increase in NIHSS caused by hemorrhage
Proportion of hemorrhagic transformation | 48 hours post-MT
All causes of death after treatment | 48 hours post-MT, 90 days post-MT

CONTACTS AND LOCATIONS:
Overall Officials: Omar Tanweer, MD, Principal Investigator — Baylor College of Medicine

REFERENCES:
- [Background] Badhiwala JH, Nassiri F, Alhazzani W, Selim MH, Farrokhyar F, Spears J, Kulkarni AV, Singh S, Alqahtani A, Rochwerg B, Alshahrani M, Murty NK, Alhazzani A, Yarascavitch B, Reddy K, Zaidat OO, Almenawer SA. Endovascular Thrombectomy for Acute Ischemic Stroke: A Meta-analysis. JAMA. 2015 Nov 3;314(17):1832-43. doi: 10.1001/jama.2015.13767. PMID 26529161
- [Background] Goyal M, Menon BK, van Zwam WH, Dippel DW, Mitchell PJ, Demchuk AM, Davalos A, Majoie CB, van der Lugt A, de Miquel MA, Donnan GA, Roos YB, Bonafe A, Jahan R, Diener HC, van den Berg LA, Levy EI, Berkhemer OA, Pereira VM, Rempel J, Millan M, Davis SM, Roy D, Thornton J, Roman LS, Ribo M, Beumer D, Stouch B, Brown S, Campbell BC, van Oostenbrugge RJ, Saver JL, Hill MD, Jovin TG; HERMES collaborators. Endovascular thrombectomy after large-vessel ischaemic stroke: a meta-analysis of individual patient data from five randomised trials. Lancet. 2016 Apr 23;387(10029):1723-31. doi: 10.1016/S0140-6736(16)00163-X. Epub 2016 Feb 18. PMID 26898852
- [Background] Kral T, Luhmann HJ, Mittmann T, Heinemann U. Role of NMDA receptors and voltage-activated calcium channels in an in vitro model of cerebral ischemia. Brain Res. 1993 May 28;612(1-2):278-88. doi: 10.1016/0006-8993(93)91673-g. PMID 8101132
- [Background] Bennion DM, Jones CH, Dang AN, Isenberg J, Graham JT, Lindblad L, Domenig O, Waters MF, Poglitsch M, Sumners C, Steckelings UM. Protective effects of the angiotensin II AT2 receptor agonist compound 21 in ischemic stroke: a nose-to-brain delivery approach. Clin Sci (Lond). 2018 Mar 15;132(5):581-593. doi: 10.1042/CS20180100. Print 2018 Mar 15. PMID 29500223
- [Background] Saver JL, Starkman S, Eckstein M, Stratton SJ, Pratt FD, Hamilton S, Conwit R, Liebeskind DS, Sung G, Kramer I, Moreau G, Goldweber R, Sanossian N; FAST-MAG Investigators and Coordinators. Prehospital use of magnesium sulfate as neuroprotection in acute stroke. N Engl J Med. 2015 Feb 5;372(6):528-36. doi: 10.1056/NEJMoa1408827. PMID 25651247
- [Background] Muir KW, Lees KR, Ford I, Davis S; Intravenous Magnesium Efficacy in Stroke (IMAGES) Study Investigators. Magnesium for acute stroke (Intravenous Magnesium Efficacy in Stroke trial): randomised controlled trial. Lancet. 2004 Feb 7;363(9407):439-45. doi: 10.1016/S0140-6736(04)15490-1. PMID 14962524
- [Background] Griauzde J, Ravindra VM, Chaudhary N, Gemmete JJ, Pandey AS. Neuroprotection for ischemic stroke in the endovascular era: A brief report on the future of intra-arterial therapy. J Clin Neurosci. 2019 Nov;69:289-291. doi: 10.1016/j.jocn.2019.08.001. Epub 2019 Aug 17. PMID 31431407
- [Background] Muir KW. Magnesium for neuroprotection in ischaemic stroke: rationale for use and evidence of effectiveness. CNS Drugs. 2001;15(12):921-30. doi: 10.2165/00023210-200115120-00002. PMID 11735612
- [Background] Muir KW. Magnesium in stroke treatment. Postgrad Med J. 2002 Nov;78(925):641-5. doi: 10.1136/pmj.78.925.641. PMID 12496316
- [Background] Lee EJ, Lee MY, Chang GL, Chen LH, Hu YL, Chen TY, Wu TS. Delayed treatment with magnesium: reduction of brain infarction and improvement of electrophysiological recovery following transient focal cerebral ischemia in rats. J Neurosurg. 2005 Jun;102(6):1085-93. doi: 10.3171/jns.2005.102.6.1085. PMID 16028768
- [Background] Marinov MB, Harbaugh KS, Hoopes PJ, Pikus HJ, Harbaugh RE. Neuroprotective effects of preischemia intraarterial magnesium sulfate in reversible focal cerebral ischemia. J Neurosurg. 1996 Jul;85(1):117-24. doi: 10.3171/jns.1996.85.1.0117. PMID 8683260
- [Background] Fraser JF, Maniskas M, Trout A, Lukins D, Parker L, Stafford WL, Alhajeri A, Roberts J, Bix GJ. Intra-arterial verapamil post-thrombectomy is feasible, safe, and neuroprotective in stroke. J Cereb Blood Flow Metab. 2017 Nov;37(11):3531-3543. doi: 10.1177/0271678X17705259. Epub 2017 Apr 21. PMID 28429604
- [Background] Feng L, Fitzsimmons BF, Young WL, Berman MF, Lin E, Aagaard BD, Duong H, Pile-Spellman J. Intraarterially administered verapamil as adjunct therapy for cerebral vasospasm: safety and 2-year experience. AJNR Am J Neuroradiol. 2002 Sep;23(8):1284-90. PMID 12223366
- [Background] Keuskamp J, Murali R, Chao KH. High-dose intraarterial verapamil in the treatment of cerebral vasospasm after aneurysmal subarachnoid hemorrhage. J Neurosurg. 2008 Mar;108(3):458-63. doi: 10.3171/JNS/2008/108/3/0458. PMID 18312091
- [Background] Albanese E, Russo A, Quiroga M, Willis RN Jr, Mericle RA, Ulm AJ. Ultrahigh-dose intraarterial infusion of verapamil through an indwelling microcatheter for medically refractory severe vasospasm: initial experience. Clinical article. J Neurosurg. 2010 Oct;113(4):913-22. doi: 10.3171/2009.9.JNS0997. PMID 19877802
- [Background] Hemmen TM, Raman R, Guluma KZ, Meyer BC, Gomes JA, Cruz-Flores S, Wijman CA, Rapp KS, Grotta JC, Lyden PD; ICTuS-L Investigators. Intravenous thrombolysis plus hypothermia for acute treatment of ischemic stroke (ICTuS-L): final results. Stroke. 2010 Oct;41(10):2265-70. doi: 10.1161/STROKEAHA.110.592295. Epub 2010 Aug 19. PMID 20724711
- [Background] Lyden P, Hemmen T, Grotta J, Rapp K, Ernstrom K, Rzesiewicz T, Parker S, Concha M, Hussain S, Agarwal S, Meyer B, Jurf J, Altafullah I, Raman R; Collaborators. Results of the ICTuS 2 Trial (Intravascular Cooling in the Treatment of Stroke 2). Stroke. 2016 Dec;47(12):2888-2895. doi: 10.1161/STROKEAHA.116.014200. Epub 2016 Nov 10. PMID 27834742
- [Background] Song W, Wu YM, Ji Z, Ji YB, Wang SN, Pan SY. Intra-carotid cold magnesium sulfate infusion induces selective cerebral hypothermia and neuroprotection in rats with transient middle cerebral artery occlusion. Neurol Sci. 2013 Apr;34(4):479-86. doi: 10.1007/s10072-012-1064-3. Epub 2012 Apr 1. PMID 22466873
- [Background] Chen J, Fredrickson V, Ding Y, Cheng H, Wang N, Ling F, Ji X. Enhanced neuroprotection by local intra-arterial infusion of human albumin solution and local hypothermia. Stroke. 2013 Jan;44(1):260-2. doi: 10.1161/STROKEAHA.112.675462. Epub 2012 Nov 27. PMID 23192754
- [Background] Shah QA, Memon MZ, Suri MF, Rodriguez GJ, Kozak OS, Taylor RA, Tummala RP, Vazquez G, Georgiadis AL, Qureshi AI. Super-selective intra-arterial magnesium sulfate in combination with nicardipine for the treatment of cerebral vasospasm in patients with subarachnoid hemorrhage. Neurocrit Care. 2009;11(2):190-8. doi: 10.1007/s12028-009-9209-9. Epub 2009 Apr 16. PMID 19370322